CLINICAL TRIAL: NCT07213921
Title: Intraoperative Dermabrasion in Mohs Surgery: A Randomized Split-Scar Trial
Brief Title: Dermabrasion in Mohs: Split-Scar Trial
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Wisconsin, Madison (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2025-0592; A534300 (Other: UW Madison); Protocol Version 3/21/25 (Other: UW Madison)
Record Dates: First submitted 2025-10-06; First posted 2025-10-09 (Actual); Last update posted 2025-10-31 (Actual); Status verified 2025-10

CONDITIONS: Wound Heal
Keywords: dermabrasion; scars
MeSH Terms: conditions — Cicatrix | interventions — Dermabrasion

STUDY DESIGN:
Intervention Model Description: This is a single center, randomized, evaluator and participant blind, split wound study.
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- A: Superior Side of the Wound (Experimental): The participant's wound will be labeled A if it is on the left or superior side of the investigator
  Interventions: Procedure: Dermabrasion
- B: Inferior Side of the Wound (Experimental): The participant's wound will be labeled B if it is on the right or inferior side of the investigator
  Interventions: Procedure: Dermabrasion

INTERVENTIONS:
Procedure: Dermabrasion — First, both sides of the wound will be sutured together with a subcutaneous (bottom) layer of stitches. Next, a predetermined, concealed randomization number will be obtained which will specify which side, A or B, will be treated with dermabrasion. An electrocautery scratch pad will be used along the wound edge of the intervention side until pin-point bleeding is achieved. This will add no additional time to the standard of care surgery time. The wound will then be closed with an epidermal (top) layer of stitches, as is the standard of care.
  Other Names: electrocautery scratch pad

SUMMARY:
The purpose of this study is to determine the potential influence of intraoperative dermabrasion on scars following Mohs Micrographic Surgery (MMS). Researchers are trying to determine if dermabrasion, a method to gently remove the top layer of your skin, is a good or bad tool to improve scar appearance after healing. The use of dermabrasion technique in this study is considered investigational. 50 participants will be enrolled and on study for up to 6 months.

DETAILED DESCRIPTION:
Primary Objective: Scar assessment at 3 months postoperatively by utilizing observer component of Patient and Observer Scar Assessment Scale (POSAS)

Secondary Objectives:

* Patient portion of POSAS
* Overall patient opinion of scar appearance
* Complication rate

ELIGIBILITY:
Inclusion Criteria:

* Able to give informed consent themselves
* Scheduled for cutaneous surgical procedure on the face or neck with predicted linear closure greater than 4 centimeters.
* Willing to return for follow up visit within the evaluation period

Exclusion Criteria:

* Patients with impaired decision-making capacity
* Significant vision or hearing impairments
* Pregnant Individuals
* Incarceration
* Wounds with predicted closure length less than 4 cm

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2025-10-23 (Actual); Primary Completion 2026-09 (Estimated); Study Completion 2026-09 (Estimated)

PRIMARY OUTCOMES:
POSAS Observer Score at 3 months post-surgery | 3 months post-surgery
  The investigators hypothesize that the side of the wound treated with intraoperative dermabrasion will have superior cosmesis as evaluated by the observer components of POSAS when evaluated at 3 months postoperatively. Two blinded reviewers will provide the POSAS Observer score which evaluates scar vascularity, pigmentation, thickness, relief, pliability, and surface area, each from 1 to 10 where higher scores indicate worse scars. Total scores are summed and range from 6-60.

SECONDARY OUTCOMES:
POSAS Patient Score at 3 months post-surgery | 3 months post-surgery
  The investigators hypothesize that the side of the wound treated with intraoperative dermabrasion will have superior cosmesis as evaluated by the patient components of POSAS when evaluated at 3 months postoperatively. The POSAS Patient score evaluates scar pain, itching, color, stiffness, thickness, and irregularity, each from 1 to 10 where higher scores indicate worse symptoms or physical scar characteristics. Total scores are summed and range from 6-60.
POSAS Overall Patient Opinion Score at 3 months post-surgery | 3 months post-surgery
  The investigators hypothesize that the side of the wound treated with intraoperative dermabrasion will have superior cosmesis as evaluated by the patient components of POSAS when evaluated at 3 months postoperatively. The POSAS overall patient opinion score ranges from 1 to 10 where higher scores indicate worse symptoms or physical scar characteristics.
Number of Complications | 3 months post-surgery

CONTACTS AND LOCATIONS:
Overall Officials: Gloria Xu, MD, PhD, Principal Investigator — UW School of Medicine and Public Health
Locations (1):
- UW Health Mohs Surgery Clinic, Madison, Wisconsin, United States

IPD SHARING:
Plan to Share IPD: Yes
Study data shared publicly (i.e.: publications, conference presentations, etc.) will be deidentified, photographs shared publicly will have participant's eyes and other identifiable features blocked to protect identity.
Supporting Information: Study Protocol, SAP, ICF